CLINICAL TRIAL: NCT00517036
Title: Omega-3 Fatty Acids for Treatment of Major Depression: Differential Effects of EPA and DHA, and Associated Biochemical and Immune Parameters
Brief Title: Omega-3 Fatty Acids for Treating Adults With Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark Rapaport, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH073765 (NIH); R01MH073765 (NIH); DATR A5-ETMA (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Depression
Keywords: Major Depression; Omega-3; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Participants will take EPA
  Interventions: Dietary Supplement: EPA omega-3 fatty acid
- B (Experimental): Participants will take DHA
  Interventions: Dietary Supplement: DHA omega-3 fatty acid
- C (Placebo Comparator): Participants will take placebo
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: EPA omega-3 fatty acid — 1 gram per day of an EPA-enriched mixture for 8 weeks
  Arms: A
Dietary Supplement: DHA omega-3 fatty acid — 1 gram per day of pure DHA for 8 weeks
  Arms: B
Dietary Supplement: Placebo comparator — 1 gram per day of an inactive substance for 8 weeks
  Arms: C

SUMMARY:
This study will test the effectiveness of two different kinds of omega-3 fatty acid dietary supplements in treating the symptoms of major depression.

DETAILED DESCRIPTION:
Major depression is a common mental disorder that affects millions of people each year. It can severely impact a person's life, causing someone to often feel sad and hopeless, as well as affect a person's sleep patterns, concentration, and energy levels. Despite the availability of numerous therapies, current treatments are not ideal for some people. Recently, some research has shown that an increase in dietary intake of polyunsaturated fatty acids (PUFAs), such as omega-3 fatty acid, might help treat depression. Eicosapentanoic acid (EPA) and docosahexanoic acid (DHA) are two common types of PUFAs high in omega-3 fatty acids and are available in low dosages in some dietary supplements. The purpose of this study is to compare the effectiveness of an EPA-enriched mixture versus pure DHA versus a placebo in treating the symptoms of major depression.

Participants in this double blind study will be randomly assigned to one of three study groups. Participants assigned to the first study group will receive capsules containing 500 mg of an EPA-enriched omega-3 fatty acid preparation. Participants assigned to the second study group will receive capsules containing 500 mg of pure DHA. Participants assigned to the third study group will receive capsules containing a placebo. The study will last approximately 9 weeks. This will include an initial screening the first week followed by an 8-week period during which all participants will take two capsules of their assigned treatment each morning. Participants will attend a total of six study visits. The initial visit will last approximately 2 hours and will include a psychiatric assessment, urine and blood collection, an electrocardiogram (EKG), and a Food Processor Questionnaire. Participants who qualify for further participation will then enter a 1-week washout period during which they will stop taking any current psychotropic medication. At the second study visit, participants will be assigned to their treatment group. Upon starting assigned treatments, participants will then return for study visits every 2 weeks to report any possible side effects and to complete standard psychiatric assessment tests. All of these study visits will take approximately 1 hour, except the last, which will take 2 hours. In addition to the psychiatric assessment and review of side effects, the final study visit will also include a physical exam and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for major depressive disorder
* A Clinical Global Impression-Severity (CGI-S) score greater than 3
* A Baseline Hamilton-D-17 (HAM-D-17) (Hamilton, 1960,1967) score of ³ 15
* Willing to use effective forms of contraception

Exclusion Criteria:

* Pregnant
* Suicidal or homicidal
* Serious or unstable medical illness, including cardiovascular, liver, kidney, respiratory, endocrine, neuralgic, or blood disease
* History of seizure disorder
* History of organic mental disorders, substance abuse, schizophrenia, schizoaffective disorder, delusional disorder, bipolar disorder, or other psychotic disorders
* History of inflammatory or auto-immune disorder (e.g., rheumatoid arthritis, multiple sclerosis, or cancer
* History of multiple adverse drug reactions or an allergy to the study drugs
* Mood-congruent or mood-incongruent psychotic features
* Current use of other psychotropic drugs
* Clinical or laboratory evidence of hypothyroidism
* Failed to respond during the course of current major depressive episode to at least one adequate antidepressant trial, defined as 6 weeks or more of treatment with 40 mg/day of citalopram (or its antidepressant equivalent)
* Received electroconvulsive therapy (ECT) within 6 months of study entry
* Currently taking supplements enriched with omega-3 fatty acids (e.g., flax seed oil) or has taken at least 1 g/day of omega-3 fatty acids
* Consuming a diet that contains more than 3g/day of omega-3 fatty acids at study entry
* Taking anticoagulants or history of a bleeding disorder
* Patients who are currently in psychotherapy that was initiated within 90 days prior to the study screening visit.
* Current infection
* Use of systematic corticosteroid or steroid antagonists or other immunosuppressant agents (e.g., cyclosporine, interferon)
* Smokes more than 10 cigarettes per day
* Taking a vitamin E supplement greater than 400 IU

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Depression rating scale score on HAM-D 17, SCID Mood Module | Both measured at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Rapaport, MD, Principal Investigator — Emory University; David Mischoulon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851
- [Derived] Mischoulon D, Nierenberg AA, Schettler PJ, Kinkead BL, Fehling K, Martinson MA, Hyman Rapaport M. A double-blind, randomized controlled clinical trial comparing eicosapentaenoic acid versus docosahexaenoic acid for depression. J Clin Psychiatry. 2015 Jan;76(1):54-61. doi: 10.4088/JCP.14m08986. PMID 25272149